CLINICAL TRIAL: NCT01224314
Title: Haemodynamic Consequences of Changing Potassium Concentrations in Haemodialysis Fluids
Brief Title: Potassium in Haemodialysis Fluids and Haemodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Regionale di Locarno (Other)
Collaborators: Fondazione Ettore Balli Locarno (Unknown)
Responsible Party: Luca Gabutti MD, Division of Nephrology, Ospedale la Carità, Via Ospedale, 6600 Locarno,Switzerland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 010010
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2007-08

CONDITIONS: Haemodialysis
Keywords: Haemodynamics; Hypotension; Potassium; Haemodialysis; Dialysis fluids
MeSH Terms: conditions — Hypotension | interventions — Dialysis Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dialysis fluid potassium high (Active Comparator): potassium concentration in the dialysis fluid 1 mmol/L higher than usual
  Interventions: Other: Changing potassium concentration in dialysis fluids
- dialysis fluid potassium low (Active Comparator): potassium concentration in the dialysis fluid 1 mmol/L lower than usual
  Interventions: Other: Changing potassium concentration in dialysis fluids

INTERVENTIONS:
Other: Changing potassium concentration in dialysis fluids — The dialysis sessions was divided into 3 tertiles, casually modulating potassium concentration in the dialysate between the value normally used K and the two cut-off points K+1 and K-1 mmol/l
  Other Names: Potassium concentrations in haemodialysis fluids

SUMMARY:
In a study published in 1995 in the American Journal of Kidney Diseases, Dolson et al demonstrated that a rapid decrease of serum potassium concentrations during haemodialysis would produce a significant increase in systolic blood pressure at the end of the session, even though there were no clear effects on intra-dialytic blood pressure. The authors defined this post-dialysis blood pressure behaviour as "rebound hypertension". Paradoxically, in animal models, other than in the context of end-stage renal disease, potassium is a vasodilator. Considering that the removal of potassium during the haemodialysis session could be theoretically modulated in profiles (as with sodium and bicarbonate), it was deemed suitable to delve deeper into this argument by studying, in detail, the (non invasive) hemodynamic repercussions of changes in the potassium concentration of the dialysate. Not being able to linearly modify the concentration, we decided to divide the dialysis session in 3 tertiles, randomising the patients to all possible dialysate sequences containing the usual concentration of potassium or two cut-off points at +1 and -1 mmol/l. Haemodynamic measurements were performed using a finger beat-to-beat monitor.

DETAILED DESCRIPTION:
INTRODUCTION:

Potassium is the most abundant cation in the body (35-40 mmol/kg in haemodialysis patients [1]), although only 2% of the pool is located extracellularly [2]. Whereas, on a short-term basis, serum potassium is regulated by the shift of potassium between the intracellular and the extracellular compartment by insulin, cathecolamines, acid-base balance, and osmolarity; kidneys are responsible for long-term potassium homeostasis [2]. Patients with end-stage renal disease are at high risk of hyperkalaemia [3-6], which may present itself as generalised weakness, paralysis, and cardiac arrhythmia [2]. Recovering potassium homeostasis is thus an important objective of dialysis. Still, considering that its location is mainly intracellular, which connects to the pharmacological concept of great distribution volume, its removal during a haemodialysis session is quantitatively modest (between 40 and 80 mmol corresponding to 1-2% of total body potassium) [1]. As a consequence, even if, in order to be suitable, potassium removal during dialysis should be equal to the amount accumulated during the inter-dialytic phase, in clinical practice the potassium concentration in the dialysate is usually adjusted with the suboptimal goal of avoiding pre-dialysis hyperkalaemia [7].

The importance of the body content and serum concentration of potassium to control blood pressure remains controversial. Epidemiological data suggest a role for potassium depletion as a co-factor in the development and severity of hypertension, while dietary potassium inversely correlates with blood pressure [8-10]. In animal models, an acute increase in serum potassium concentration produces vasodilatation mediated by the vascular endothelium; the opposite effect is observed if it decreases [11,12]. In haemodialysis, the extent of the difference between serum potassium and the potassium concentration in the dialysis fluid is directly correlated to an increase in blood pressure at the end of the dialysis session, producing what has been named "rebound hypertension" [1]. In this same study no significant changes in blood pressure were found during the dialysis.

In haemodialysis the nephrologists are faced with sudden changes in blood pressure and haemodynamic fragility phases that have a multi-factorial origin; ultrafiltration, decrease in osmolarity with imbalance and correction of metabolic acidosis play a predominant role [13-19]. Despite this, and thanks to some artifices, with particular reference to calcium concentration in the dialysate [15], dialysate temperature [20] and ultrafiltration and sodium concentration profiles [18,21-24], pressure stability is guaranteed as a general rule. Some electrolytes, particularly sodium and bicarbonate, can be modulated in profiles with the purpose of better respecting the gap in osmolarity or concentration that is established during the haemodialysis session, but their haemodynamic effect still remains controversial [20,22,24].

Serum potassium is an electrolyte whose concentration - in order to guarantee a negative balance - varies rapidly and significantly during dialysis, frequently resulting in going from pre-dialysis hyperpotassaemia to intra-dialysis hypopotassaemia. As mentioned above, in Dolson's study [1], differences in dialyses blood pressure were not found between the groups treated with dialysates containing 1, 2 or 3 mmol/l of potassium, but at the end of the dialyses those patients treated with the lower potassium concentrations showed what was called a "rebound hypertension".

With the purpose of better characterising this phenomenon, we redesigned the study dividing the dialysis session into 3 phases (in fact, clinical practice suggests that the haemodynamic pattern at the beginning, intermediate and final phases of the dialysis are not the same) and programming for each a more or less sharp drop in serum potassium concentration, respecting in the meantime the need to remove the amount of potassium that usually keeps the patient in steady-state. Using a crossover research model, we divide the dialysis session in 3 tertiles where the potassium concentration in the dialysate was modulated between the usual concentration for the study subject and two cut-off points at +1 e -1 mmol/l respectively. To complete the information provided by blood pressure, haemodynamics were measured in a non-invasive manner using a finger beat-to-beat monitor.

The primary end point was the difference in haemodynamic parameters between the extremes in potassium concentration of the dialysate, while the incidence of hypotension during dialysis was considered a secondary end point.

METHODS:

Twenty-four chronic haemodialysis patients (13 male and 11 female) were enrolled in the study. Each patient was dialysed for 3 to 4 hours and 30 minutes three times a week and was clinically stable and without intercurrent illnesses. Using a single blind crossover design, patients were randomised in the six dialysate potassium sequences of the study. Each dialysis session was divided into three equal parts (tertiles): during one part the potassium concentration of the dialysate was the same as the one usually prescribed to the patient, whereas during the other two parts it was either increased or reduced by 1 mmol/L. The 6 different permutations were repeated twice, so that each patient underwent 12 dialysis sessions during the study (see Table 1 for sequence details).

The haemodialyses were performed using a 4008 H machine, equipped with a cartridge of bicarbonate Bibag©, and a high flux single use polysulfone membrane, all from Fresenius Medical Care (Bad Homburg, Germany). The prescribed dialyser effective surface area, dialysis fluid conductibility, dialysate temperature and composition (with the exception of potassium concentration), effective blood flow, and dry weight were recorded at the enrolment in the study and were then left unchanged. The medications of the patients were also left unchanged. Serum potassium and patient weight were measured at the beginning and at the end of each dialysis session. Blood samples were taken from the arterial limb of the shunt.

Kt/V was used to quantify haemodialysis adequacy and was calculated using a second generation single-pool Daugirdas formula (Kt/V = -ln(R-0.03) + [(4-3.5 x R) x (UF/W)], where R = post-dialysis BUN/pre-dialysis BUN, UF = net ultrafiltration, W = weight, K= dialyzer clearance of urea, t= dialysis time, and V= patient's total body water.

The incidence of hypotension episodes (defined as a systolic blood pressure < 90 mmHg) was recorded.

Systolic and diastolic blood pressures, heart rate, stroke volumes (integrated mean of the flow waveform between the current upstroke and the dicrotic notch) and total peripheral resistances (ratio of mean arterial pressure to stroke volume multiplied by heart rate) were evaluated at the beginning of the session and then every 30 minutes using a Finometer© finger beat-to-beat monitor (Finapres Medical Systems BV, Arnhem, The Netherlands). Finometer© measures finger blood pressure noninvasively on a beat-to-beat basis and gives waveform measurements similar to intra-arterial recordings.

Mean blood pressure (BPmean) was calculated using the following formula: BPmean=(BPsyst+2BPdias)/3, where BPsyst and BPdias are systolic and diastolic blood pressure, respectively.

The fluid loss as a function of the time was considered to be constant during the dialysis session and was recorded as total ultrafiltration.

Statistical analyses were performed using the SAS System (Statistical Analysis System). Comparisons between body weight, potassium concentration and haemodynamic parameters were done first with an ANOVA and followed, if significant by a paired t-test performed between the mean values obtained in each patient with each modality. To improve the probability of showing significant differences, the haemodynamic parameters within the tertiles were compared against the dialysate potassium concentration cut-off points (-1 vs. +1 mmol/l). Percentages were compared using a Fisher Exact test. In all cases, a P ≤ 0.05 was considered statistically significant; P was expressed as ns (not significant) and as significant (P ≤0.05).

REFERENCES:

See Citations

ELIGIBILITY:
Inclusion Criteria:

* chronic haemodialysis patients
* dialysed 3 to 4 hours three times a week
* clinically stable and without intercurrent illnesses

Exclusion Criteria:

* intercurrent illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
haemodynamic consequences of dialysate potassium concentration | 4 weeks
  difference in haemodynamic parameters between the extremes in potassium concentration of the dialysate

SECONDARY OUTCOMES:
incidence of hypotension | 4 weeks
  incidence of hypotension during dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gabutti, MD, Principal Investigator — Ospedale Regionale di Locarno
Locations (1):
- Ospedale Regionale di Locarno, Locarno, Canton Ticino, Switzerland

REFERENCES:
- [Background] Dolson GM, Ellis KJ, Bernardo MV, Prakash R, Adrogue HJ. Acute decreases in serum potassium augment blood pressure. Am J Kidney Dis. 1995 Aug;26(2):321-6. doi: 10.1016/0272-6386(95)90652-5. PMID 7645536
- [Background] Rastegar A, Soleimani M. Hypokalaemia and hyperkalaemia. Postgrad Med J. 2001 Dec;77(914):759-64. doi: 10.1136/pmj.77.914.759. PMID 11723313
- [Background] Bia MJ, DeFronzo RA. Extrarenal potassium homeostasis. Am J Physiol. 1981 Apr;240(4):F257-68. doi: 10.1152/ajprenal.1981.240.4.F257. PMID 6111930
- [Background] Fernandez J, Oster JR, Perez GO. Impaired extrarenal disposal of an acute oral potassium load in patients with endstage renal disease on chronic hemodialysis. Miner Electrolyte Metab. 1986;12(2):125-9. PMID 3960016
- [Background] Perez GO, Pelleya R, Oster JR, Kem DC, Vaamonde CA. Blunted kaliuresis after an acute potassium load in patients with chronic renal failure. Kidney Int. 1983 Nov;24(5):656-62. doi: 10.1038/ki.1983.208. PMID 6663988
- [Background] Musso CG. Potassium metabolism in patients with chronic kidney disease. Part II: patients on dialysis (stage 5). Int Urol Nephrol. 2004;36(3):469-72. doi: 10.1007/s11255-004-6194-y. PMID 15783126
- [Background] Locatelli F, Covic A, Chazot C, Leunissen K, Luno J, Yaqoob M. Optimal composition of the dialysate, with emphasis on its influence on blood pressure. Nephrol Dial Transplant. 2004 Apr;19(4):785-96. doi: 10.1093/ndt/gfh102. PMID 15031331
- [Background] Morris RC Jr, Sebastian A, Forman A, Tanaka M, Schmidlin O. Normotensive salt sensitivity: effects of race and dietary potassium. Hypertension. 1999 Jan;33(1):18-23. doi: 10.1161/01.hyp.33.1.18. PMID 9931076
- [Background] Stamler J, Rose G, Elliott P, Dyer A, Marmot M, Kesteloot H, Stamler R. Findings of the International Cooperative INTERSALT Study. Hypertension. 1991 Jan;17(1 Suppl):I9-15. doi: 10.1161/01.hyp.17.1_suppl.i9. PMID 1987018
- [Background] Whelton PK, He J, Cutler JA, Brancati FL, Appel LJ, Follmann D, Klag MJ. Effects of oral potassium on blood pressure. Meta-analysis of randomized controlled clinical trials. JAMA. 1997 May 28;277(20):1624-32. doi: 10.1001/jama.1997.03540440058033. PMID 9168293
- [Background] Amberg GC, Bonev AD, Rossow CF, Nelson MT, Santana LF. Modulation of the molecular composition of large conductance, Ca(2+) activated K(+) channels in vascular smooth muscle during hypertension. J Clin Invest. 2003 Sep;112(5):717-24. doi: 10.1172/JCI18684. PMID 12952920
- [Background] Haddy FJ, Vanhoutte PM, Feletou M. Role of potassium in regulating blood flow and blood pressure. Am J Physiol Regul Integr Comp Physiol. 2006 Mar;290(3):R546-52. doi: 10.1152/ajpregu.00491.2005. PMID 16467502
- [Background] Rodrigo F, Shideman J, McHugh R, Buselmeier T, Kjellstrand C. Osmolality changes during hemodialysis. Natural history, clinical correlations, and influence of dialysate glucose and intravenous mannitol. Ann Intern Med. 1977 May;86(5):554-61. doi: 10.7326/0003-4819-86-5-554. PMID 851303
- [Background] van der Sande FM, Kooman JP, Leunissen KM. Intradialytic hypotension--new concepts on an old problem. Nephrol Dial Transplant. 2000 Nov;15(11):1746-8. doi: 10.1093/ndt/15.11.1746. No abstract available. PMID 11071958
- [Background] Gabutti L, Bianchi G, Soldini D, Marone C, Burnier M. Haemodynamic consequences of changing bicarbonate and calcium concentrations in haemodialysis fluids. Nephrol Dial Transplant. 2009 Mar;24(3):973-81. doi: 10.1093/ndt/gfn541. Epub 2008 Oct 8. PMID 18842671
- [Background] Gabutti L, Ferrari N, Giudici G, Mombelli G, Marone C. Unexpected haemodynamic instability associated with standard bicarbonate haemodialysis. Nephrol Dial Transplant. 2003 Nov;18(11):2369-76. doi: 10.1093/ndt/gfg383. PMID 14551368
- [Background] Sulowicz W, Radziszewski A. Dialysis induced hypotension--a serious clinical problem in renal replacement therapy. Med Pregl. 2007;60 Suppl 2:14-20. PMID 18928150
- [Background] Leunissen KM, Kooman JP, van Kuijk W, van der Sande F, Luik AJ, van Hooff JP. Preventing haemodynamic instability in patients at risk for intra-dialytic hypotension. Nephrol Dial Transplant. 1996;11 Suppl 2:11-5. doi: 10.1093/ndt/11.supp2.11. PMID 8803987
- [Background] Selby NM, McIntyre CW. A systematic review of the clinical effects of reducing dialysate fluid temperature. Nephrol Dial Transplant. 2006 Jul;21(7):1883-98. doi: 10.1093/ndt/gfl126. Epub 2006 Apr 6. PMID 16601075
- [Background] van Kuijk WH, Wirtz JJ, Grave W, de Heer F, Menheere PP, van Hooff JP, Leunissen KM. Vascular reactivity during combined ultrafiltration-haemodialysis: influence of dialysate sodium. Nephrol Dial Transplant. 1996 Feb;11(2):323-8. doi: 10.1093/oxfordjournals.ndt.a027261. PMID 8671787
- [Background] Kim MJ, Song Jh, Kim Ga, Lim Hj, Lee Sw. Optimization of dialysate sodium in sodium profiling haemodialysis. Nephrology (Carlton). 2003 Oct;8 Suppl:S16-22. doi: 10.1046/j.1440-1797.8.s.2.x. PMID 15012686
- [Background] Stefanidis I, Stiller S, Ikonomov V, Mann H. Sodium and body fluid homeostasis in profiling hemodialysis treatment. Int J Artif Organs. 2002 May;25(5):421-8. doi: 10.1177/039139880202500512. PMID 12074340
- [Background] Stiller S, Bonnie-Schorn E, Grassmann A, Uhlenbusch-Korwer I, Mann H. A critical review of sodium profiling for hemodialysis. Semin Dial. 2001 Sep-Oct;14(5):337-47. doi: 10.1046/j.1525-139x.2001.00086.x. PMID 11679103
- [Derived] Gabutti L, Salvade I, Lucchini B, Soldini D, Burnier M. Haemodynamic consequences of changing potassium concentrations in haemodialysis fluids. BMC Nephrol. 2011 Apr 6;12:14. doi: 10.1186/1471-2369-12-14. PMID 21470404